CLINICAL TRIAL: NCT01415895
Title: A Proof-of-Concept, Randomized, Double-Blind and Placebo Controlled Clinical Trial With Naltrexone and Clonidine Combination (ATNC05) Compared With Placebo in the Treatment of Chronic Back Pain
Brief Title: Naltrexone and Clonidine Combination (ATNC05) in the Treatment of Chronic Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annette C. Toledano MD (Industry)
Responsible Party: Sponsor-Investigator, Annette C. Toledano MD, Sponsor/Investigator, Allodynic Therapeutics, Inc
Organization: Allodynic Therapeutics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT110491
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Back Pain; Lower Back Pain; Cervical Pain
Keywords: back pain; cervical pain; neuropathic pain; radicular pain
MeSH Terms: conditions — Back Pain; Low Back Pain; Neck Pain; Neuralgia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATNC05 - a study drug capsule (Experimental): Naltrexone and Clonidine Combination (ATNC05)
  Interventions: Drug: Naltrexone and Clonidine Combination
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Naltrexone and Clonidine Combination — subjects will receive 1 study drug capsule by mouth twice daily for 3 weeks, followed by 1 capsule in the morning for 3 days.
  Other Names: ATNC05
  Arms: ATNC05 - a study drug capsule
Drug: placebo — subjects will receive 1 placebo capsule by mouth twice daily for 3 weeks, followed by 1 capsule in the morning for 3 days.
  Arms: placebo

SUMMARY:
The study includes back pain of the cervical, thoracic, and the lumbar regions.

ELIGIBILITY:
Inclusion Criteria:

The subject has chronic back pain for > 3 months in the lumbar, thoracic or cervical regions.

The average pain intensity scale during the screening week is 4/10 - 8/10 (On an 11-point Numeric Pain Intensity Scale with 0 = no pain and 10 = worst pain imaginable).

The subject has not taken Opioid medications 7 days prior to initiation of study drug.

The subject has a heart rate of 60bpm or above and/or systolic blood pressure 90 or above.

The subject is willing to refrain from using NSAIDS, Acetaminophen or muscle relaxants, unless for rescue, for the duration of the study The subject is willing to refrain from using Opioid medications and excessive alcohol for the duration of the study.

The subject is able to read, understand and follow the study instructions, including completion of questionnaires at home.

The subject must sign an informed consent document indicating willingness to participate.

If the subject is a female, she must be post-menopausal, not currently pregnant or nursing. A female of child bearing potential should be using a reliable contraception method during the course of the study.

Exclusion Criteria:

The subject has a positive urine drug screen. The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.

The subject has any significant deviations from normal in physical examination, electrocardiogram (ECG), Echocardiogram or clinical laboratory tests, as evaluated by the investigator.

The subject has a history of an allergic reaction to the components of the study drug.

The subject has acute back or cervical pain. The subject has muscular back or cervical pain. The subject has back or cervical pain other than chronic Radicular pain.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Brief Pain Inventory 24-hour Pain Scores for average pain (Question #5) | baseline to week 3
  The Brief Pain Inventory is a self-reported medical questionnaire used to measure pain over the past 24-hours - worst pain (Question 3), least pain (Question 4), average pain (Question 5), right now pain (Question 6) and at night pain (Question 7). The score ranges from 0 to 10 (0 - no pain) (10 - intolerable pain).

SECONDARY OUTCOMES:
Change from Baseline in Brief Pain Inventory 24-hour assessment of interference in function (Questions 9a - 9i). | baseline to week 1, week 2 and week 3
  BPI Interference; questions 9a - 9i - measures a self-reported assessment of the interference in function because of pain in past 24 hours in general activity, mood, walking ability, normal work, relationship with other people, sleep quality, enjoyment of life, standing ability and sitting ability. Interference scores: 0 (does not interfere) to 10 (completely interferes).
Change From Baseline in Brief Pain Inventory 24-hour subject's Global Impression of Improvement (Question 8) | baseline to week 1, week 2 and week 3
  The Brief Pain Inventory question 8 measures the subject's perception of how much relief he has received at the time of assessment compared with before the start of the study drug. The score is measured in percentage 0% (no relief) to100% (complete relief).
Change From Baseline in the subject's Global Assessment of Treatment Satisfaction today | baseline to week 1, week 2 and week 3
  A self-reported scale that measures Treatment Satisfaction today in (0-10, 0 - none, 10 - most satisfied)
Change from Baseline in the subject's perception of Ability to Tolerate the study drug and the severity of side effects today. | baseline to week 1, week 2 and week 3
  A self-reported scale that measures the ability to tolerate the study drug and the severity of side effects today in (0-10, 0 - No side effects, 10 - intolerable side effects)
Change From Baseline in Oswestry Disability Index and Neck Disability composite scores(ODI), to Week 1, Week 2, and Week 3 | baseline to week 1, week 2 and week 3
  The Oswestry Low Back Pain Disability Questionnaire (Oswestry Disability Index) and Neck Disability composite assesses pain-related disability in persons with low back pain (LBP) and neck pain. The score is recorded in percentage of disability.
Change From Baseline in Roland Morris Disability Questionnaire composite scores(ODI), to Week 1, Week 2, and Week 3 | baseline to week 1, week 2 and week 3
  The Roland Morris Disability Questionnaire consists of 24 statements and the subject is instructed to put a mark next to each appropriate statement. The total score ranges from 0 (no disability) to 24 (severe disability).
Change From Baseline in Vital Signs - systolic blood pressure, diastolic blood pressure, pulse rate and body mass index to Week 1, Week 2, and Week 3. | baseline to week 1, week 2 and week 3
Change from Baseline to week 3 in Laboratory Assessments - Alkaline Phosphatase, Alanine Transaminase - ALT (SGPT), Aspartate transaminase - AST(SGOT), Bilirubin, Total, Serum Creatinine, Blood Urea Nitrogen, Serum Chloride, Potassium, HCO3 | baseline to week 1, week 2 and week 3
Change from Baseline in the investigator's Clinical Global Impression - Severity scale (CGI-S) to Week 1, Week 2, week 3 . | baseline to week 1, week 2 and week 3
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the investigator to rate the severity of the subject's back pain at the time of assessment, relative to the investigator's past experience. Considering total clinical experience, the subject is assessed on severity of back pain at the time of rating 1, normal; 2, borderline; 3, mild; 4, moderate; 5, marked; 6, severe; or 7, extreme.
Change from Baseline in The investigator's Clinical Global Impression - Improvement scale (CGI-I) to Week 1, Week 2, week 3 | baseline to week 1, week 2 and week 3
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale, the investigator will rate how much the patient's back pain has improved or worsened relative to a baseline state at the beginning of the study and rate as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Change from Baseline in the subject's answer to the question, "Are you better off today then the time before starting the study drug?, yes/no, by what percentage? | baseline to week 1, week 2 and week 3
  Answer, yes/no and by 0%-100% (0%-not at all better, 100% - very much better off
Change From Baseline in the subject's answer to the question " Have you been more / less active in the past 24 hrs, comparing to the period before initiating the study drug, please rate in %. | baseline to week 1, week 2 and week 3
  The subjects answer, one of the following choices, - 150%, -100%, -50%, - 25%, 0% - same activity level, +25%, +50%, +100%, +150%
Subject's response to the question, "Have you responded to the treatment?" | baseline to week 1, week 2 and week 3
  Subject's answer yes/no.
Subject's Global Assessment of Disease Activity Improved / No Change | baseline to week 1, week 2 and week 3
  The Subject answer either Improved or No Change.
Subject's Global Evaluation of Study Medication. | baseline to week 1, week 2 and week 3
  The subject chooses, 1 - Excellent, 2 - Very Good, 3 - Good, 4 - Fair, 5 - Poor
The Subject's Satisfaction with Pain Relief, 0 - 10. | baseline to week 1, week 2 and week 3
  The subject answers on a scale of 0-10, (0 - not satisfied, 10 - very satisfied).
The Subject's Satisfaction with Moving, Standing, Walking and Bending Ability Scale, 0-10. | baseline to week 1, week 2 and week 3.
  The subjects answers on a scale of 0-10, (0 - not satisfied, 10 - very satisfied)
Change from Baseline in Brief Pain Inventory 24-hour Pain Scores for worst pain, least pain, right now pain and night pain (Questions 3,4,6 & 7) | baseline to week 1, week 2 and week 3
  The Brief Pain Inventory is a self-reported medical questionnaire used to measure pain over the past 24-hours - worst pain (Question 3), least pain (Question 4), average pain (Question 5), right now pain (Question 6) and at night pain (Question 7). The score ranges from 0 to 10 (0 - no pain) (10 - intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Annette C Toledano, MD, Principal Investigator — Allodynic Therapeutics, Inc
Locations (1):
- Annette C. Toledano MD, North Miami, Florida, United States